CLINICAL TRIAL: NCT03053141
Title: RHythmia mAPping and Signal acquisitiOn for Data analYsis (RHAPSODY)
Acronym: RHAPSODY
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 91087667
Record Dates: First submitted 2016-05-24; First posted 2017-02-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrythmias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- All Subjects: All subjects are included in this cohort and are treated with the Rhythmia Mapping System
  Interventions: Device: Rhythmia Mapping System

INTERVENTIONS:
Device: Rhythmia Mapping System — The Rhythmia Mapping System is a 3D electro-anatomical mapping system.

SUMMARY:
The objective of the RHAPSODY study is to evaluate the performance of new software features in subjects undergoing standard of care catheter-based endocardial mapping for atrial or ventricular tachyarrhythmias using a commercial Rhythmia Mapping System. Results from this study will be used to guide development and refinement of new software features that may be implemented in future commercial software releases.

DETAILED DESCRIPTION:
The Rhythmia Mapping System is designed for electroanatomical mapping in catheter ablation procedures by optimizing the need for speed and accuracy. The system is able to simultaneously acquire data from multiple electrodes. In addition, based on user-defined criteria, the system is able to efficiently acquire data over multiple cardiac beats. When used in conjunction with the Rhythmia Mapping Catheter, the system is able to acquire up to hundreds of points per minute leading to fast and detailed map creation.

Since its market release, physicians and users have gained experience with the Boston Scientific Rhythmia Mapping System in the human clinical setting. Improvements to the first generation system are in development and include new and improved software features and mapping algorithms to enhance the clinical operation. These new and improved software features and algorithms require leveraging clinical use data as part of the development and iteration process.

This study will evaluate the performance of potential next-generation software features in a low-risk clinical environment by streaming raw signals from a commercial Rhythmia Workstation during standard of care cardiac mapping and ablation treatments for tachyarrhythmias, specifically atrial fibrillation, atrial tachycardias, and ventricular tachycardia. The data will be evaluated on a parallel investigational Rhythmia Workstation using prototype software features. These next-generation software features and algorithms will not be available to the physician during the case and will therefore have no diagnostic or therapeutic impact on the clinical case.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above, or above legal age and willing and capable of giving informed consent specific to national law
2. Scheduled for standard of care catheter-based endocardial mapping for atrial or ventricular tachyarrhythmias using a commercial Rhythmia Mapping System.

Exclusion Criteria:

1. Prothrombotic or bleeding tendency due to coagulopathy or blood dyscrasia
2. Inability to tolerate heparin therapy (e.g. heparin induced thrombocytopenia, allergy, etc.)
3. Prosthetic or stenotic valves in the chamber where the intended mapping will occur, or in the path of the catheter access route
4. Active systemic infection or sepsis
5. Hemodynamic instability or shock at baseline precluding ablation in the assessment of the investigator.
6. Presence of intracardiac thrombus, tumor, or other abnormality which precludes catheter introduction
7. Women who are pregnant or lactating
8. Cardiac surgery within the past 90 days
9. Acute myocardial infarction within 3 months
10. Stable/unstable angina or ongoing myocardial ischemia
11. Subjects with an active heart failure decompensation
12. Long QT Syndrome, Brugada Syndrome, or Torsade de Pointes
13. Congenital heart disease with or without corrective surgery that would complicate a mapping procedure
14. Subjects having untreatable allergy to contrast media
15. Vascular pathology or tortuosity precluding standard vascular access techniques
16. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for standard of care catheter-based endocardial mapping for atrial or ventricular tachyarrhythmias using a commercial Rhythmia Mapping System.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Physician Feedback on Software Performance | 1 day- Procedure
  Physician Feedback on Software Performance

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H McElderry, MD, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Lukes Idaho Cardiology Associates, Boise, Idaho
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Catholic Medical Center, Manchester, New Hampshire
  - Valley Hospital, Ridgewood, New Jersey
- Fondazione Centro San Raffaele, Milan, MI, Italy
- Centre Hospitalier Princesse Grace, Monaco, Monaco